CLINICAL TRIAL: NCT04113941
Title: A Randomized, Double-Blind, Placebo-controlled, Multi-center, Phase 3 Study to Evaluate the Efficacy and Safety of MEDITOXIN® in Subject With Idiopathic Overactive Bladder
Brief Title: Clinical Trial to Evaluate the Efficacy and Safety of MEDITOXIN® in Subject With Idiopathic Overactive Bladder
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Medy-Tox (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MT01-KR17OAB302
Record Dates: First submitted 2019-07-01; First posted 2019-10-03 (Actual); Last update posted 2020-07-28 (Actual); Status verified 2020-07

CONDITIONS: Overactive Bladder
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neuronox® (Experimental): Neuronox® total 100U, inject 5U/0.5mL per site, 20 sites
  Interventions: Drug: Neuronox
- Placebo (Placebo Comparator): Normal saline, same volume with Experimental arm
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Neuronox — intradetrusor injection
  Other Names: Meditoxin
  Arms: Neuronox®
Drug: Placebo — intradetrusor injection
  Arms: Placebo

SUMMARY:
This study is for patients who have idiopathic overactive bladder symptoms. This study will evaluate efficacy and safety of Neuronox® against placebo.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects aged above 20
* Patient with overactive bladder symptoms lasting at least 6 months

Exclusion Criteria:

* Patient with a history of surgery or a disease that may affect bladder function.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2019-08-23 (Actual); Primary Completion 2020-04-15 (Actual); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
The change in the daily average UI (Urinary Incontinence) episodes | 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Konkuk University Hospital, Seoul, South Korea